CLINICAL TRIAL: NCT04207502
Title: Integrating Systematic Data of Geriatric Medicine to Explore the Solution for Health Aging
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Chang Gung University (Other)
Responsible Party: Sponsor
Other Study IDs: CORPG3J0371; 201900702A3 (Other: Chang Gung Medical Foundation)
Record Dates: First submitted 2019-11-26; First posted 2019-12-23 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-09

CONDITIONS: Sleep Disturbance; Cognitive Change; Aging
Keywords: dementia; depression; brain structure; system biology
MeSH Terms: conditions — Parasomnias; Dementia; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood, urine, and stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project aims to build up the comprehensive database of geriatric medicine for local Taiwanese.

DETAILED DESCRIPTION:
This project is the pilot for the basis of establishing the schema of database and efficient procedures including subject recruitment, specimen collection, management, and measurement of samples obtained from multiple sources. We will focus on deciphering the correlation of sleep quality and the integrity of brain structure by integrating the holistic health data, socio-demographic characteristics, MRI, wearable technique, and laboratory technology including clinical lab, genotyping, metabolomics, gut microbiome, to unravel the clinical feature of which the age will effect on the frequency of sleep disturbance. This project will not only systematically study the aging effect on the sleep quality and brain structure integrity, but pave the way for exploring a variety of aging-related indications.

ELIGIBILITY:
Inclusion Criteria:

* Participants of annual health checkup conducted by either Taipei city or Chang Gung Health and Culture Village.
* aged ≧ 60 years old.
* have medical record in Chang Gung Memorial Hospital.
* resided in the Taiwan area over 180 days in past one year.

Exclusion Criteria:

* Participants with the medical history of severe organ disorders, severe autoimmune disease, or cancer under treatment.
* Contraindications or previously failure for receiving brain computerized tomography or magnetic resonance imaging scan.
* Participants who had receive outpatient clinic follow-ups with diseases that may affect the cognitive evaluation or presentation.
* Depression with ongoing diagnosis and treatment, suicide idea or suicide behavior in the past 6 months.
* Difficulty in communication or disabilities

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 subjects with aged over 60 years old participated in annual health checkup conducted by either Taipei city or Chang Gung Health and Culture Village.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
The brain volume of local Taiwanese aged over 60 years old | one hour
  Measure the volume of cerebrum, cerebellum, and skin of skull (unit in mm3) by magnetic resonance imaging (MRI)
The monitoring of sleep-related events of local Taiwanese aged over 60 years old | one night
  Measure the sleep stages (unit in minute), apnea-hypopnea index (unit in counts/hour), and respiratory events by polysomnography

SECONDARY OUTCOMES:
The actigraphy of local Taiwanese aged over 60 years old | two weeks
  Measure the circadian rhythm (unit in minute) by Actiwatch
The neurocognitive questionnaire of local Taiwanese aged over 60 years old | one day
  Measure the neurocognitive condition and sleep quality as assessed by GDS-15, UCLA-LS, HAM-A, HAM-D, AES, TSII, CTQ, AD8, MMSE, ECog, CERAD-NAB, PSQI, ESS, SOS, and STOP-Bang
The gut microbiota of local Taiwanese aged over 60 years old | one day
  Assess the gut bacterial diversity and profile by stool analysis
The metabolism of local Taiwanese aged over 60 years old | one day
  Measure the metabolites as biomarkers by urine and blood analysis
The polysomnographic recording for elderly with obstructive sleep apnea (OSA) | three months
  Subjects with OSA will undergo continuous positive airway pressure (CPAP) and evaluate the improvement rate (unit in percent) by polysomnography and sleepiness questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: JI-TSENG FANG, M.D., Study Chair — Chang Gung Memorial Hospital; NING-HUNG CHEN, M.D., Principal Investigator — Chang Gung Memorial Hospital; GENG-HAO LIU, M.D., Principal Investigator — Chang Gung Memorial Hospital; JUNG LUNG HSU, M.D., Principal Investigator — Chang Gung Memorial Hospital; SHWU-HUA LEE, M.D., Principal Investigator — Chang Gung Memorial Hospital; CHIH-MING LIN, M.D., Principal Investigator — Chang Gung Memorial Hospital; CHUNG-HAO LIN, M.D., Principal Investigator — Chang Gung Memorial Hospital; CHENG HONG TOH, M.D., Principal Investigator — Chang Gung Memorial Hospital; CHENG-HSUN CHIU, M.D., Principal Investigator — Chang Gung Memorial Hospital; MEI-LING CHENG, Ph.D., Principal Investigator — Chang Gung University
Locations (2):
- Taiwan (2):
  - Taipei Chang Gung Memorial Hospital, Taipei
  - Chang Gung Health and Culture Village, Taoyuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu GH, Huang YH, Yuan TC, Chen YP, Hsu JL, Lee SH, Lin CM, Toh CH, Fang JT, Lin SW, Chuang LP, Chen NH. Associations of Wearable-Measured Sleep and Physical Activity With Memory Performance in Older Adults: Cross-Sectional Study With Actigraphy and MRI. JMIR Aging. 2025 Dec 9;8:e80584. doi: 10.2196/80584. PMID 41258815